CLINICAL TRIAL: NCT06418217
Title: 3 Months Semi-supervised Exercise Intervention for Patients With Hip Abductor Tendon Pathology (HATP): A Prospective Clinical Cohort Study
Brief Title: Exercise and Patient Education for Patients With Lateral Hip Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jeppe Lange (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor-Investigator, Jeppe Lange, MD, PhD, Horsens Hospital
Organization: Horsens Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-16-02-180-24
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Gluteal Tendinitis; Greater Trochanteric Pain Syndrome; Hip and Thigh Injury; Rupture of Hip Abductor Tendon (Disorder)
Keywords: Exercise; Patient education; Lateral Hip Pain; Rehabilitation
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physiotherapist-led exercise (Experimental): Physiotherapy-led exercise of patients with lateral hip pain
  Interventions: Procedure: Exercise and Patient Education

INTERVENTIONS:
Procedure: Exercise and Patient Education — Patients will undergo a 12-week physiotherapist-led exercise program consisting of 8 supervised sessions and home-based training in between.
  Patients will keep training diaries, where each session is tracked in regards of completed repetitions and pain before and after the sessions. Each session will consist of four exercises.

SUMMARY:
This prospective cohort trial will investigate a progressive exercise protocol and patient education for patients with hip abductor tendon pathology. The primary outcome is patient reported pain measured by the revised Copenhagen Hip And Groin Outcome Score (HAGOS), that will be conducted at baseline and at a 12 week follow-up.

DETAILED DESCRIPTION:
This study protocol describes an interventional pragmatic prospective single-group cohort study, where the primary endpoint is change in hip pain measured with the revised HAGOS pain subscale following a 12 week intervention. Throughout the 12 weeks, eight physiotherapist-led exercise sessions will take place at Horsens Regional Hospital (HRH). Further, at the sessions at HRH patient education will be performed by the supervising physiotherapist. The first supervised sessions will be performed in continuation of the baseline assessment. The patients will be instructed to do the exercises daily at home in the time period between the physiotherapist-led sessions.

The primary aim is to investigate changes in patient-reported hip pain based on the subscale "pain" from the revised Copenhagen Hip And Groin Outcome Score (HAGOS) from baseline to 12 week follow-up.

It is hypothesized that the revised HAGOS pain score will improve from baseline to 12 week follow-up.

Secondarily explorative subgroup analyses regarding whether patients with different MRI findings, pain profiles, age, sex and body mass index (BMI) respond differently to the intervention, will be performed.

All outcomes conducted will be published. That is, patient-reported outcomes, muscle strength, functional capacity and adherence to the exercise protocol.

A full study protocol will be published and made available.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* MRI verified HATP
* Lateral hip pain duration > 6 months
* Ability to read and understand Danish.

Exclusion Criteria:

* Corticosteroid injection in the affected hip joint within the last six weeks prior to the intervention
* Previous bone-related surgery to the affected hip,
* Signs of bilateral HATP
* X-ray verified hip osteoarthritis
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes in patient-reported pain measured with the revised Copenhagen Hip And Groin Outcome Score (HAGOS) (continuous data) | From baseline to 3 months follow-up. The outcome is also conducted at 6-week follow-up.
  The subscale "pain" on HAGOS measures the patients perception of hip and/or groin pain. It consist of ten items. A score from 0 to 100 is calculated, where a higher score is indicating lower pain.

SECONDARY OUTCOMES:
Changes in patient-reported symptoms measured with the revised Copenhagen Hip And Groin Outcome Score (HAGOS) (continuous data) | From baseline to 3 months follow-up. The outcome is also conducted at 6-week follow-up.
  The subscale "symptoms" on HAGOS measures the patients perception of hip and/or groin pain. It consist of seven items. A score from 0 to 100 is calculated, where a higher score is indicating lower symptoms.
Changes in patient-reported physical function in daily living (ADL) measured with the revised Copenhagen Hip And Groin Outcome Score (HAGOS) (continuous data) | From baseline to 3 months follow-up. The outcome is also conducted at 6-week follow-up.
  The subscale "ADL" on HAGOS measures the patients perception of hip and/or groin pain. It consist of five items. A score from 0 to 100 is calculated, where a higher score is indicating higher function.
Changes in patient-reported physical function in sport and recreational activities (sport/recreation) measured with the revised Copenhagen Hip And Groin Outcome Score (HAGOS) (continuous data) | From baseline to 3 months follow-up. The outcome is also conducted at 6-week follow-up.
  The subscale "sport/recreation" on HAGOS measures the patients perception of hip and/or groin pain. It consist of eight items. A score from 0 to 100 is calculated, where a higher score is indicating higher function.
Changes in patient-reported participation in physical activities (PA) measured with the revised Copenhagen Hip And Groin Outcome Score (HAGOS) (continuous data) | From baseline to 3 months follow-up. The outcome is also conducted at 6-week follow-up.
  The subscale "PA" on HAGOS measures the patients perception of hip and/or groin pain. It consist of two items. A score from 0 to 100 is calculated, where a higher score is indicating higher ability to participate in physical activity.
Changes in patient-reported quality of life (QOL) measured with the revised Copenhagen Hip And Groin Outcome Score (HAGOS) (continuous data) | From baseline to 3 months follow-up. The outcome is also conducted at 6-week follow-up.
  The subscale "QOL" on HAGOS measures the patients perception of hip and/or groin pain. It consist of five items. A score from 0 to 100 is calculated, where a higher score is indicating higher quality of life.
Changes in the patient-reported outcome measure Oxford Hip Score (continuous data) | From baseline to 3 months follow-up. The outcome is also conducted at 6-week follow-up.
  Oxford Hip Score (OHS), which consists of 12items. OHS is developed and validated for patients undergoing total hip replacements to access pain and function. It is a composite score ranging from 0 (worst) to 48 (best).
Changes in the patient-reported outcome measure EQ-5D-5L (continuous data) | From baseline to 3 months follow-up. The outcome is also conducted at 6-week follow-up.
  European Questionnaire-5 Dimensions (EQ-5D-5L and EQ-VAS) consists of five items and a visual analogue score (VAS), a vertical line on which the patients score their perception of their overall health from 0 to 100 (worst to best)
Global Rating of Change (GRoC) | The outcome is conducted at 6-week and 3-months follow-up.
  GRoC consists of a 11-point scale, where the patient rates the perceived overall change of the hip condition from "very much better" to "very much worse" . Responses on GRoC will be considered successful if patients scored "moderately better" to "very much better". Global improvement will be measured as the percentage of successful reports.
Lateral hip pain on a numerical pain rating scale (NRS) | From baseline to 3 months follow-up. The outcome is also conducted at 6-week follow-up.
  Participants rate their pain on a scale from 0 (no pain) to 10 (worst imaginable). Participants will rate their average pain for the past 7 days during rest, at the beginning of activity, during activity, 2 hours after activity and the worst lateral hip pain.
Changes in the patient-reported outcome measure The Victorian Institute of Sport Assessment-Gluteal Questionnaire (VISA-G) (continuous data) | From baseline to 3 months follow-up. The outcome is also conducted at 6-week follow-up.
  The Victorian Institute of Sport Assessment-Gluteal Questionnaire (VISA-G) is validated for patients with gluteal tendinopathy and measures the severity of disability related to the condition. VISA-G consist of eight items and appraise the pain in relation to gluteal tendinopathy by a score from 0-100, where a higher score will indicate lower pain and less disability.
Changes of maximal isometric hip abduction muscle strength (continuous data) | From baseline to 3 months follow-up. The outcome is also conducted at 6-week follow-up.
  Maximal isometric hip abduction strength test measures the maximal voluntary isometric contraction in supine position. The strength will be measured using a fixed dynamometer. Strength will be conducted in Newton, but will be normalised according to the lever arm and body weight, and will be reported as Nm/kg bodyweight.
Changes of maximal isometric hip adduction muscle strength (continuous data) | From baseline to 3 months follow-up. The outcome is also conducted at 6-week follow-up.
  Maximal isometric hip adduction strength test measures the maximal voluntary isometric contraction in supine position. The strength will be measured using a fixed dynamometer. Strength will be conducted in Newton, but will be normalised according to the lever arm and body weight, and will be reported as Nm/kg bodyweight.
Changes of maximal isometric hip flexion muscle strength (continuous data) | From baseline to 3 months follow-up. The outcome is also conducted at 6-week follow-up.
  Maximal isometric hip flexion strength test measures the maximal voluntary isometric contraction in sitting position. The strength will be measured using a fixed dynamometer. Strength will be conducted in Newton, but will be normalised according to the lever arm and body weight, and will be reported as Nm/kg bodyweight.
Changes of maximal isometric hip extension muscle strength (continuous data) | From baseline to 3 months follow-up. The outcome is also conducted at 6-week follow-up.
  Maximal isometric hip extension strength test measures the maximal voluntary isometric contraction in prone position. The strength will be measured using a fixed dynamometer. Strength will be conducted in Newton, but will be normalised according to the lever arm and body weight, and will be reported as Nm/kg bodyweight.
Changes of the number of repetitions of a 30 second sit to stand test (continuous data) | From baseline to 3 months follow-up. The outcome is also conducted at 6-week follow-up.
  Number of repetitions (sits to stand) performed during 30 seconds on a chair with a seat height of 45 cm.

OTHER OUTCOMES:
Adherence to the exercise program. | From baseline to 3 months follow-up.
  The adherence will be calculated as the proportion of completed exercise sessions in relation to the planned exercise sessions. A high adherence will be defined as completion of 75% or more of the planned exercises sessions (both supervised and home-based), medium adherence with completion of 50-74%, and low adherence with completion of less than 50%.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Høgsholt, PT, PhD.st., Principal Investigator — Horsens Regional Hospital; Aarhus University; Jeppe Lange, MD, PhD, Study Director — Horsens Regional Hospital; Aarhus University; Signe Kierkegaard-Brøchner, PhD, Study Chair — Regionshospitalet Horsens; Kristian Thorborg, PhD, Study Chair — Copenhagen University Hospital, Hvidovre; Marie Bagger Bohn, MD, PhD, Study Chair — Regionshospitalet Horsens
Locations (1):
- Horsens Regional Hospital, Horsens, Horsens, Denmark

IPD SHARING:
Plan to Share IPD: Yes
What data will be shared: All quantitative individual participant data collected during the trial, after deidentification, and according to current Danish Data Protection Regulation and GDPR.
  With whom will data be shared: Researchers who provide a methodologically sound proposal.
  For what types of analyses: To achieve aims in the approved proposal. The abovementioned is based on Data Sharing Statements for Clinical Trial: A Requirement of the ICMJE located at: https://www.icmje.org/news-and-editorials/data_sharing_june_2017.pdf
Supporting Information: Study Protocol
Time Frame: Immediately following publication and ending 5 years following primary article publication.
Access Criteria: Proposals should be directed to mathhg@rm.dk. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Hogsholt M, Kierkegaard-Brochner S, Lange J, Thorborg K, Bohn MB. Physiotherapist-led education and exercise for patients with MRI-verified hip abductor tendon pathology: a protocol for a prospective cohort study. BMJ Open. 2025 Sep 11;15(9):e106517. doi: 10.1136/bmjopen-2025-106517. PMID 40940047